

# **CONSENT FORM and HIPAA Authorization**

### Study Title: Folks-At-Risk for Interstitial Lung Disease (FAR-ILD)

Study number: IRB-AAAR1916

Anticipated number of subjects: 800

Patel, MD; Da Zhang MD; Belinda D'Souza MD; Mary Principal Investigator: Christine Kim Garcia MD on Anderson MD; Matthew Baldwin MD; Keith Brenner PhD; Sean Fedyna MD; Claire McGroder MD; Nina Salvatore MD; Anjali Saqi MD; and David Goldstein MD; William Bulman MD; Wellington Cardoso, MD, behalf of the following investigators: Michaela

email: mac2463@cumc.columbia.edu; Tel: 212-342-Contact person: Mohammad "Atif" Choudhury; 4551 or 646-641-3521.

#### Introduction

The purpose of this form is to give you information to help you decide if you want to take part in a research study. This consent and HIPAA authorization form includes information about:

- Why the study is being done;
- The things that you will be asked to do if you are in the study;
  - Any known risks involved;
- Any potential benefit;
- Options, other than taking part in this study, that you have; and
  - The way your health information will be used and shared for research purposes.

The principal investigator (the lead researcher for this the study team. Take all the time you need to decide whether you want to take part in this research study. questions about the study, please ask a member of discuss this study with you. If at any time you have involved in this project), or a study coordinator will project, a co-investigator (another researcher

the 'What is Involved in This Study?' section of this The purpose of this research is described below in consent form.

## What information is on this form?

from you. Please take the time to read this form. We research study. Participation is voluntary; you do not ike to use information about you and how we would need to decide whether you want to take part in the This form explains why we are doing this study and participate in it. It also describes the way we would We are asking you to take part in a research study. ike to use the blood and tissue samples we obtain research study. If at any time you have questions about this for or the research study, please ask a member of the study team. Take all the time you what you will be asked to do if you choose to will also talk with you about taking part in this have to participate if you do not want to.

## Why is this study being done?

understanding of the cause of interstitial lung disease been asked to participate in the study either because (ILD), including the use of genetic testing. You have specific genes or genetic variants. We are collecting well as from individuals at risk for developing ILD. If Medical Center (CUMC) and will be studied with the and possibly confirm associations between ILD and goal of identifying causes and contributors to these you have been diagnosed with ILD or because you results of the genetic tests being performed to find you agree to participate, your samples and clinical individuals who have been diagnosed with ILD as DNA/RNA samples and clinical information from information will be stored at Columbia University are at risk for developing ILD. We will study the The purpose of this study is to gain a better conditions.

will undergo a CAT scan of their chest to assess their with ILD. Participants over the age of 40 years of age age will undergo breathing tests to assess their lung lung health. Participants over the age of 35 years of health in adults who have another family member At-Risk Family Members. We are assessing lung health.

history. Participants who have received a diagnosis of chest to assess their lung health. At-risk smokers are have been diagnosed with bronchiectasis will not be adults. Participants will undergo a CAT scan of their At-Risk Smokers. We are assessing lung health for chronic obstructive pulmonary disease "COPD: are eligible to participate if they are 50 year of age and eligible to participate. However, participants who above with a minimum of 30 pack-year smoking eligible to participate

age will undergo a CAT scan of their chest to assess At-Risk COVID-19 Survivors. We are assessing lung pneumonia. Participants over the age of 21 years of health of adults who have survived a COVID-19 their lung health. Participants will also undergo breathing tests.

control if you are a household contact of someone Controls. You might be asked to participate as a who is recruited to participate in this study.

### What will I be asked to do if I choose to be in this study?

Patients with ILD:

- We will collect medical information and CAT scan images from your medical record.
  - We will collect a sample of blood.
    - We may collect a nasal swab.
- If you have undergone a biopsy of your lung, we may use some of the lung tissue for research.
  - We may ask you to return to see us each year.
- The study will follow-up with you for up to 20 years. Patients with ILD who are not being treated at New
  - York Presbyterian/Columbia University Medical Center will be asked to sign a medical release form, the information obtained will be used for research purposes only.

At-Risk Family Members and Survivors of COVID-19 lung disease:

- We will ask you to come to New York
- Presbyterian/Columbia University Medical Center. A doctor will ask you questions about your health and perform a partial physical examination.
  - We will collect a sample of blood
    - We may collect a nasal swab.



- We will ask you to perform two breathing tests (called pulmonary function tests):
- A "spirometry" test to measure the flow of air in and out of your lungs. This will require you to breathe in hard and deep and blow out over a period of time. At least 3 and as many as 6 exhalation efforts will be necessary for this test.
   A "diffusing capacity" test to measure how well your lungs exchange oxygen and carbon dioxide. You breathe in and hold your breath for 10 seconds, then rapidly blow it out.
  - We will ask you to walk for 6 minutes in a hallway walking test.
    - We will ask you to undergo a CAT scan of your chest, which involves radiation.
- We may invite you to undergo a bronchoscopy (described below) to obtain small pieces of your lung for research tests.

At-Risk Participants with Smoking History:

- We will ask you questions regarding your smoking history.
- We will collect a sample of blood.
  - We may collect a nasal swab.
- We will ask you to undergo a CAT scan of the chest, which involves radiation. If you have undergone a CAT scan of the chest within the past year, we will ask you to either provide us with a copy of the scan or sign a medical release form so that the research staff can obtain a copy of the
- We may also invite you to undergo pulmonary function testing as well.
- We may invite you to undergo bronchoscopy (described below) to obtain small pieces of your lung for research tests.

#### Controls:

- We will ask questions about your health and collect information about you. We will specifically ask if you have been diagnosed with a lung ailment.
  - We will collect a samples of blood and may collect a nasal swab. These samples may be used for genetic testing and results may be returned to you (see below).
    - You will not be asked to undergo bronchoscopy.

Bronchoscopy:

Presbyterian. If you undergo a bronchoscopy, you will lungs to limit the amount of cough and discomfort you the tip. The doctor will be able to see the inside of the "bronchoscope" through your nose or mouth and then cells, and saline (salt water) washings of the inside of pregnant. You will have an "IV" (intravenous) catheter Depending on your test results, we may invite you in placed so that medications can be given to you. The study doctor will give you medications that will make general anesthesia as a routine part of this research long, thing, flexible medical device with a camera on bronchoscopy. If you are a woman, we may ask you (lidocaine) into your nose, throat, and airways in the into the airways of your lungs. A bronchoscope is a to undergo a biopsy of your lung using a procedure need to have blood drawn again for "routine" blood the lungs. A bronchoscopy is a medical procedure called a bronchoscopy, to obtain lung tissue, lung performed by a doctor. The bronchoscopy will be airways of your lungs, take pictures, and will also for a urine sample to determine whether you are you sleepy ("sedation"), but you will not receive study. The doctor will put numbing medication performed in a procedure room at New York perform the following procedures using the might experience. The doctor will place a tests to make sure it is safe to perform a bronchoscope:

- 1. The doctor will take biopsies of your lung tissue. This means that the doctor will remove small pieces of your lung tissue (the airsacs and airways of your lungs) using cutting devices for research purposes. This tissue will be used for research.
- The doctor will use a small brush to collect cells from the inside lining of your nose and airways. These cells will be used for research.
- The doctor will put salt water (saline) into your lung to wash out any cells that may be there.
   Some of the salt water will be removed by the bronchoscope and used for research.

If there are unexpected findings in your lungs during the bronchoscopy, the study doctor may perform additional procedures (such as more biopsies) to try to find out what these unexpected findings are. You

and your doctor will be informed of the results of any additional procedures for unexpected findings.

After the bronchoscopy you will have at least one chest x-ray to make sure the lungs look healthy. A second chest x-ray is sometimes needed. If you undergo bronchoscopy, we will call you one month later to check your health status.

Please write your initials next to the choice you make below:

(initial) yes, I agree to bronchoscopy with biopsy, fluoroscopy and a chest x-ray, which include radiation.

(initial) no, I do not agree to bronchoscopy with biopsy, fluoroscopy and a chest x-ray, which include radiation.

For all Subjects:

Blood samples.

We will ask you to give a blood sample of up to 25mL (about 5 teaspoons) at enrollment and up to 45mL at follow-up visits. The blood will be drawn (taken) using a needle in a vein and sent to be stored in our research laboratory for future genetic testing. If a blood sample cannot be obtained, you will be asked to provide a saliva sample or buccal (cheek swab) sample. Samples collected for this study will be used to extract DNA and RNA. Some of your blood samples will also be stored in Dr. Garcia's laboratory for future research.

Follow-up evaluations.

We may ask you to return to see us each year, whether you undergo a bronchoscopy or not. The study will follow-up with you for up to 20 years.

Future Use of Data/Specimens

We would like to store the data and biological samples that you agreed to provide as part of this study and use them for future research. They will be stored at CUMC indefinitely either with the researchers on this study or in a central storage facility called a repository. By signing this consent, you agree that your samples can be stored at CUMC indefinitely for future research. Your samples and data will be labeled with a code number that the researchers on this study will be able to link to you. You also agree that Your samples Real Dec Steped in



entities, that may not yet be identified, for research of ILD or other conditions. If your data and samples are shared with researchers who are not researchers on your data and samples may be used in the future by have access to the repository will not be able to link them to you. By signing this consent, you agree that de-identified form, which mean that individuals who removed from your data and samples OR that your who will use them will not have the key to the code Any future testing or research using your data and information, products, tests and treatments having data and samples are coded and the researchers samples may lead to the development and use of compensation that may result from these tests or this study, they will only be given in de-identified researchers at other institutions or commercial identifying information have been permanently form. This means that your name and other commercial value. You will not receive any Dr. Garcia, other CUMC researchers, and treatments.

You can change your mind regarding storage and future use of your samples at any time. Please see the Contact section of the consent form for further information.

access to the data. This means that researchers who request access to the data must promise that they will Because our research is funded by various sponsors, by the database rules, report any data breeches and the researchers on this study. We would only submit protect the data, only share that data as is permitted genetic data to a data storehouse not maintained by so that individuals who have access to the database we have taken steps to de-identify your data, it may you through your genetic information in combination with data from other public sources. We believe that not seek to identify any individuals from the data. If will not be able to link the data to you. Even though storehouse it will be submitted in de-identified form be possible that someone might be able to identify your data to a storehouse that permits controlled your data is submitted to an outside public data we may be required to submit your clinical and Long-term storage of your data. this is unlikely to happen.

# What are the risks of participating in this study? There may be slight pain or bruising due to the blood draw. We will use only skilled individuals to obtain blood from you.

Pulmonary Function Tests may cause lightheadedness, dizziness, and/or syncope.

Even without your name and other identifiers, your genetic information is unique to you. There is a potential risk that someone will identify you from your genetic information or learn something about you by looking at your genetic information; this risk may increase in the future as technologies advance and more researchers study your genetic information. These risks may also affect members of your family. You should discuss your participation in this study with your family and ask the study doctor about any questions or concerns you may have.

The Genetic Information Non-discrimination Act (GINA) is a federal law that prevents insurance companies from using your genetic information to deny health insurance coverage. The law also prevents employers from getting or using genetic information for employment-related decisions. However, the law does not prevent companies that provide life insurance, disability insurance or longterm care insurance from using genetic information.

Current genetic testing is not an exact science, and you should be aware that the genetic testing being done in this study is considered research testing. As with all research, it is possible that although the tests gives us information that we think may be important, we will not know what all of it means. Thus, it is possible that the meaning of the information you are given may change over time as additional research is conducted.

The genetic research may identify genetic changes that may require additional testing to evaluate. This could result in anxiety, uncertainty and additional expenses that may or may not be covered by your insurance. The genetic research may identify serious, untreatable genetic conditions. Such a finding can result in unexpected psychological trauma, both for you and your family. The detection of such a condition could also affect the health or health care

needs of your siblings, children or other close relatives. Because we cannot say with certainty how information derived from the genetic research could be used in the future, this study may involve risks that are currently unforeseeable.

#### Radiation

Radiation is an energy that is all around us. It is in the Radiation and the risks of receiving radiation are hard energy used in X-rays and some other types of scans air, water, food, and ground. This is called natural radiation. Radiation is also made by humans. It is in our lifetime. You should always carefully think about to measure. Experts on radiation agree that there is some risk because radiation exposure adds up over Tomography, or PET, scans) is known as radiation. examinations or treatments. The "effective dose" of radiation is measured in millisievert (mSv) units. On receives about 3.1 mSv/year from natural radiation. how much radiation you will receive from medical People receive about 2.2 mSv/year from flying in examinations or treatments such as X-rays. The the average, each person in the United States (such as bone density and Positron Emission our buildings and homes. It is also in medical airplanes.

This research study includes exposure to radiation. This radiation exposure is not required for your medical care and is for research purposes only. The radiation exposure is necessary to obtain the research information desired. If you have had X-rays in the past or have been exposed in other ways to radiation, or if you think that you might be pregnant, you must tell the investigator before you agree to be in the study.

In this study, you will receive radiation from a chest CT scan. If you are invited to participate in the bronchoscopy sub-study you will also receive radiation from fluoroscopy and a chest x-ray.

The procedure involving radiation from the chest CT scan in this research study will expose you to a very small amount (up to 15 mSv) of radiation. There may be an increase in the chances of your developing cancer many years after this study. The additional risk from this research study is less than 0.3%.



Columbia University IRB IRB-AAAR1916 (Y05M00)
IRB-Approval Date: 11/18/2020 For use until: 11/17/2021

If you are invited to participate in the bronchoscopy sub-study, this research study will expose you to an additional very small amount (1.3 mSv) of radiation from fluoroscopy and a chest X-ray. In this case, the total amount of radiation is 16.3 mSv and the total risk is 0.33%.

At these very low levels, scientists are uncertain as to the actual risk from research and there may be no

In addition, the procedures involving radiation in this research study (e.g. fluoroscopy) might increase the possibility of skin injury, hair loss and/or cataracts. Skin injuries seldom occur and are usually limited to a small area of reddening of the skin surface that was irradiated. They rarely result in an ulcer. If hair loss occurs, it is usually temporary, but could be permanent. Cataracts occur rarely and appear many years after the exposure of the eyes to large doses of radiation.

## **Bronchoscopy and Biopsy**

There are risks if you undergo a bronchoscopy and biopsy. Up to 1 out of 50 people who undergo bronchoscopy for a medical reason can expect to have a complication. When complications occur, they are typically minor and are related either to the procedure itself or to medications used during the procedure.

Sedation that you receive during the bronchoscopy can cause low blood pressure, low oxygen levels, high carbon dioxide levels, nausea, vomiting (which can lead to pneumonia).

Topical anesthetics ("numbing medication") can cause seizures, heart rhythm abnormalities, and can affect the ability of your blood to carry oxygen.

Bronchoscopy (along with washings and brushings of the airways) can often cause nasal discomfort, sore throat, chest pain, low-grade fevers, low oxygen levels (requiring the use of oxygen), and pneumonia. Less common complications of bronchoscopy include asthma-like reactions with wheezing, low oxygen levels, fainting, injury or swelling of the voice box in the throat, injury to the airways (bronchi) in the lung,

or serious infections. Rarely, the bronchoscopy equipment could malfunction and damage you.

A lung biopsy performed during bronchoscopy increases the risk of the procedure. About 1 out of 30 people will have bleeding and 1 out of 50 will have a collapse of their lung (a "pneumothorax"). Almost all bleeding episodes are mild and resolve spontaneously or with medications. Collapsed lungs are also typically mild and can be treated with oxygen or with a small or large tube placed between the ribs to drain the air. Rarely, one or more life-threatening complications can occur including severe bleeding, severe collapse of the lung, severe abnormal heart rhythms, cardiac arrest (when the heart stops beating), or respiratory failure (when the lungs stop working).

Death is extremely rare, but can occur in up to 1 out of 10,000 bronchoscopies. You should know that we are aware of one healthy person who died after undergoing a bronchoscopy for research purposes. This occurred in 1996 at another hospital not affiliated with our hospital.

## Pregnancy/breastfeeding risks

Taking part in this study while you are pregnant could cause harm to your fetus. If you are breastfeeding, taking part in this study could cause harm to your baby. You must not take part in this study if you are pregnant or breastfeeding.

### Loss of confidentiality

A risk of taking part in this study is the possibility of a loss of confidentiality. Loss of confidentiality includes having your personal information shared with someone who is not on the study team and was not supposed to see or know about your information. The study team plans to protect your confidentiality. Their plans for keeping your information private are described in the 'confidentiality' section of this consent form.

### Incidental Findings

Although the imaging (CAT scan) you will have in this study is being undertaken for research purposes only, it is possible that doctors may notice something that could be important to your health, such as a nodule in your lungs. Although not likely, it is possible that the

doctors may notice something that may be very serious and could immediately affect your life. If so, we will contact you to explain what was observed. If you so desire, we will also talk with your private physician. If you do not have a private physician, we will refer you to an appropriate clinic for follow-up. It will be your choice whether to proceed with additional tests and/or treatments to evaluate what we observed, and you or your insurer will be responsible for these costs.

# Are there benefits to taking part in this study?

If you agree to take part in the study, and choose to receive results, there may be direct medical benefit to you.

If your CAT scan or biopsy identifies a medical condition, it is possible that your health could be improved by treating that condition.

If a genetic predisposition for a medical condition is found, knowing this information may help determine how to manage your medical care. We hope that in the future, information learned from this study will benefit other people with similar findings.

However, if the sequencing does not find information that would affect your medical care or well being, there may not be any direct benefit to you. The knowledge gained may increase our understanding of genetic testing and results of genetic tests, and help patients in the future.

#### Confidentiality

To help us protect your privacy, we have obtained a Certificate of Confidentiality from the National Institutes of Health. The researchers can use this Certificate to legally refuse to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings. For example, if there is a court subpoena, the researchers will use the certificate to resist any demands for information that would identify you, with the following exceptions listed below.

- The Certificate cannot be used to resist a demand for information from personnel of the United States federal or state government agency sponsoring the project and that will be used for auditing or program Columbia University IRB

IRB-AAAR1916 (Y05M00) IRB Approval Date: 11/18/2020 For use until: 11/17/2021

σ information that must be disclosed in order to meet Administration (FDA). You should understand that involvement in this research. If an insurer, medical care provider, or other person obtains your written researchers will not use the Certificate to withhold Certificate of Confidentiality does not prevent you consent to receive research information, then the the requirements of the federal Food and Drug releasing information about yourself or your or a member of your family from voluntarily evaluation of agency funded projects or for that information.

regarding matters such as child abuse and neglect, The Certificate of Confidentiality will not be used to prevent disclosure to state or local authorities or harm to self or others.

however, complete confidentiality cannot be promise. identify you by name will be kept confidential. We will such as a stolen computer may occur, although it is Any information collected during this study that can Despite all of our efforts, unanticipated problems do everything we can to keep your data secure, highly unlikely.

protected health information and information collected If you choose to take part in this study, you are giving us the authorization (i.e. your permission) to use the during the research that can identify you. The health be considered sensitive. The research study will not research may include medical information that may collect HIV test results, history of drug or alcohol information that we may collect and use for this abuse, or mental health information.

involved in your care that is needed for this research Information about you may be obtained from any hospital, doctor, and other health care provider

name, address, telephone number or any other direct New York-Presbyterian Hospital will not include your Any research information that is shared with people outside of Columbia University Medical Center and identified unless disclosure of the information is required by law or you have authorized the disclosure.

research file that links your name to the code number responses, and health information will be assigned a and authorized study staff will have access to the file. code number, and separated from your name or any password-protected computer. Only the investigator other information that could identify you. The Your data, biological samples, questionnaire will be kept in a locked file cabinet and on a

record (EMR) system, which will be shared with Weill Cornell Medical Center, and New York-Presbyterian recently implemented a new electronic medical Columbia University Irving Medical Center has Hospital and its affiliated institutions.

personnel from these institutions. Study monitors and records in this system can be viewed by authorized others who provide oversight of the study may also Your participation in this research study will be documented in our new EMR system. Medical need to access this record. The following individuals and/or agencies will be able to look at, copy, use, and share your research information.

- medical professionals who may be evaluating the York-Presbyterian Hospital study staff and other Center, Weill Cornell Medical Center, and New - The investigator, Columbia University Medical study.
- Staff and authorities from Columbia University, and New York-Presbyterian Hospital, including the Institutional Review Board (IRB)
  - ('OHRP') and the United States Food and Drug The Office of Human Research Protections Administration ('FDA')
- National Institute of Health

information does not have an expiration (ending) Your authorization to use and share your health date

α participating in a study), federal privacy laws may not Once your health information has been disclosed to third party (for example, a pharmaceutical company longer protect it from further disclosure.

this consent and authorization at any time and for any You may change your mind and revoke (take back)

reason. To revoke this consent and authorization, you must contact the Principal Investigator,

650 West 168th Street, BB9-903D Dr. Christine Garcia

disclose the information they have already collected. taking part in the research. Also, even if you revoke this consent and authorization, the researchers and the sponsor (if applicable) may continue to use and authorization, you will not be allowed to continue However, if you revoke your consent and New York, NY, 10032

What other options are there? You may choose not to take part in this research study.

# What if I get hurt while I am on the study?

or harm to you. In the event of an injury resulting from appropriate medical care and inform the study doctor. Taking part in this research study may result in injury In the event of an emergency you should go to an your participation in this study, you should seek emergency room.

through the New York-Presbyterian Hospital (NYPH), a Columbia doctor, or any other health provider, you participating in the study and receive medical care receive. All or part of your bill may be paid by your will be sent a bill for whatever medical care you If you are injured or harmed as a result of health insurance.

non-medical care costs that might occur as a result of Columbia University and the New York-Presbyterian Hospital (NYPH) are not offering to pay you for pain, worry, lost income, the cost of your medical care or your taking parting this study. However, you do not waive any of your legal rights in signing this form.

### Will I get compensated?

Patient(s) with ILD:

- You will not receive any payment or compensation for taking part in this study.

### Individuals At-Risk for ILD:

If you are eligible for compensation, you will receive - You will receive \$100 for completing the initial your compensation in the form of a gift card.

Columbia University IRB IRB-AAR(1916 (Y05M00) IRB Approval Date: 11/18/2020 For use until: 11/17/2021 resear¢⊓



- You will receive \$50 for completing the annual follow-up research visit.
  - You will receive \$100 for completing the bronchoscopy portion of the study.

-You will receive \$25 for completing the visit.

# Will I incur costs if I take part in this study?

You will incur no costs to be in this study. You will not including genetic tests that may be recommended by research. However, you or your insurance company be charged for the costs of confirming in a clinical your physician as a result of information received will be responsible for any additional clinical test, laboratory any genetic findings to be used in

## Do I have to be in the study?

any time. Your choice will not affect the treatment you decide not to take part in or stop being in the study at receive from doctors and staff at Columbia University Medical Center and New York-Presbyterian Hospital. Taking part in this study is your choice. You can

updated information about your health, or to provide a clarify information that you have provided, or to obtain Why might researchers want to contact me in the consent form you are giving us permission to contact contact you in the future. They may want to obtain a new sample of blood or saliva or cheek swab, or to future? The researchers of this study may want to preliminary result from this study. By signing this you in the future for research purposes.

which could be important to you or a family member's us if you want to know about this genetic test result or It is possible that in the future, a genetic test could be health. Knowing this information could have risks. For make it difficult to get certain types of insurance. If Dr. notified about genetic test results, the research study example, it may make you anxious. Or, if the results team will contact you. You will have the option to tell done on your stored samples that may give results, Garcia and the researchers believe that the genetic are discovered by insurance companies, it could test results are important and if you agree to be

# What are my rights if I take part in this study?

affect your access to health care at CUMC or NYPH. any time. Your choice will not involve any penalty or decide not to take part or stop being in the study at Taking part in this study is your choice. You can loss of benefits to which are entitled and will not

consent form if you decide to withdraw from the study your biological samples are they have been de-linked specify in your written notice if you want your unused databases, and, if you have given your permission to from identifying information or deposited in scientific that your samples and/or data will not be included in on our ability to exclude your information or remove any future analyses. However, there are limitations information removed from all CUMC databases so biological samples destroyed and your identifying researchers listed in the Contact section of this contacted by the researchers. You will need to do so, used or shared with other researchers. before it is finished and no longer want to be You will need to notify in writing one of the

# Whom may I call if I have questions?

If you have any questions about this research study, you may contact:

Dr. Christine Kim Garcia by e-mail at ckg2116@cumc.columbia.edu

research participant, or if you have a concern about If you have any questions about your rights as a this study, you may contact the office below.

Columbia University Medical Center Human Research Protection Office E-mail: irboffice@columbia.edu 154 Haven Avenue, 1st Floor Telephone: (212) 305-5883 Institutional Review Board New York, NY 10032

organized to protect the rights and welfare of human An Institutional Review Board is a committee subjects involved in research.

study can be found on the Columbia University IRB website at: http://www.cumc.columbia.edu/dept/irb More information about taking part in a research

## Some Background on Genes

the genome that includes only the DNA that is directly Your entire unique genetic material, made up of DNA, is known as a 'genome.' An 'exome' is the portion of responsible for telling cells how to make the correct parts, or proteins, to function properly.

contained in most of the cells that make up the body's brief explanations. Please let us know, at any point, if 'gene.' Abnormalities in the information in a gene can We would like you to be well informed about genetic tissues. DNA carries the instructions for your body's lead to disease. Your entire unique genetic material, inheritance of many human traits, such as hair and research, and for that reason we have, next, a few cells how to make the correct parts, or proteins, to 'exome' is the portion of the genome that includes only the DNA that is directly responsible for telling determines a specific function of a cell is called a understand. DNA is the material that governs the development and functions. A piece of DNA that eye color or the risk of some diseases. DNA is you want or need more information in order to made up of DNA, is known as a 'genome' An function properly.

about unexpected diseases. Because WES and WGS are more comprehensive than other genetic tests, it is their relationship to interstitial lung diseases. Genetic Because WES and WGS examine a larger portion of can cause disease. WGS searches through all of the did not. WES and WGS may also reveal information searches through the exome for DNA variations that tests that may be developed in the future. WES and perform whole exome sequencing but other genetic research is evolving rapidly. We expect that we will WGS are very detailed types of genetic tests. WES the genetic material than traditional tests, they may ests in addition to, or in the place of, whole exome be able to find causes of disease where other tests biological samples to identify variants and consider What are Whole Exome Sequencing and Whole sequencing (WES) or whole genome sequencing (WGS) may be performed, including new genetic Genome Sequencing? We are requesting your genome, including areas outside of the exome. permission to perform genetic testing on your



particularly important that you understand what is involved. The study coordinator will tell you more about WES and WGS. You may also wish to obtain professional genetic counseling prior to signing this consent form. If genetic variants are found, the IGM will make a genetic counselor available to you, your family members and/or your physician in the event that you have additional questions regarding the results of your testing at no cost. However, you or your insurance provider will be responsible for all costs related to your medical care, including clinic visits and medical procedures recommended to you as a consequence of study results.

## Will I get a genetic test result?

Genetic information generated by and clinical information recorded as a part of this research study will be analyzed by study investigators in order to identify genetic causes for interstitial lung diseases. Although the goal of the study is to generate as much genetic data as is possible, there is no guarantee that your sample or data will be analyzed. It is highly unlikely that we will discover genetic variants that have such strong effects that they would be considered to be the cause of your disorder therefore you will probably receive no results from this study. However, it is possible that the cause of your ILD might be determined by the research team.

It is possible that a genetic test will give results that the study team believes are linked to some or all features of your disease. It is also possible that a genetic test may predict that you are at increased risk for developing ILD in the future. Knowing this information could have risks. For example, it may make you anxious. Or, if the results are discovered by insurance companies, it could make it difficult to get some kinds of insurance.

Dr. Garcia and the researchers are giving you the option to tell us if you want to be notified about genetic test results. If a genetic test result is found that may impact your medical care and if you want to be notified about genetic test results, you will be contacted that a result has been found that requires further testing. If you are a patient of one of the physicians conducting this study, the research staff will facilitate a referral to a clinic or physician who can

order the confirmatory test. Please note that this consent form contains space for you to name a physician you wish to be involved in disclosing results of the confirmatory genetic test you.

You might need to provide an additional blood sample for confirmatory genetic testing. You might be offered genetic counseling as part of this study, or pursue genetic counseling outside of this study. The cost of confirmatory genetic testing is provided by this study.

If you do not have ILD, a positive test might mean that you may be predisposed (i.e., more likely to develop) heart/lung disease. If this is the case, your physician may order additional medical tests. The cost of these additional medical tests are not covered by this study.

If you do have ILD, it is important for you to understand that this study may not identify a cause for your condition because:

- Your ILD is not due to a genetic cause
- A genetic variant exists, but based on current knowledge, it cannot be determined whether it is related to your ILD. In these cases, you will not be informed of any results. Your sample may be used, however, for future tests.

If there is a positive test result, you may want to undergo further independent testing and/or consultation with specialist physicians and/or genetic counselors. Genetic counseling is provided through the study; however independent testing and consultation with a medical geneticist or other medical specialist is not. You should be aware that insurance companies sometimes use information from genetic testing to deny coverage to applicants (see information on GINA above).

Please choose and initial one of the options below to tell us if you want to know about genetic test results now and in the future.

(initial) Yes, please contact me if information is found in studies of my genetic material that would be important to me or my family's personal health. Please note that I wish to include the physician listed below to be involved in disclosing results of

confirmatory genetic testing to me. The following physician: \_\_\_\_ (print name) practicing in \_\_\_\_ (city, state) should be involved in disclosing results of confirmatory genetic testing to me.

(initial) No, don't contact me about information found in studies of my genetic material.

### Statement of Consent

I voluntarily consent to participate in the study. I have read this consent and HIPAA authorization form which includes information about the nature and the purpose of the study, as well as a description of study procedures.

I have discussed the study with the investigator or study staff, have had the opportunity to ask questions and have received satisfactory answers. The explanation I have been given has mentioned both the possible risks and benefits to participating in the study and the alternatives to participation.

I understand that I am free to not participate in the study or to withdraw at any time. My decision to not participate, or to withdraw from the study will not affect my future care or status with this investigator.

I understand that I will receive a copy of this signed and dated consent form and HIPAA authorization. By signing and dating this consent form, I have not waived any of the legal rights that I would have if I were not a participant in the study.

#### Study Participant Print Name

Signature \_\_\_\_\_

Date & Time

Person Obtaining Consent Print Name

Signature \_\_

Date & Time # Columbia

